CLINICAL TRIAL: NCT02244593
Title: FAST MRI Study in Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Jean Seely, Dr. Jean Seely, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OHSN-REB 20140103-01H
Record Dates: First submitted 2014-06-06; First posted 2014-09-19 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: breast cancer survivors; FAST MRI; mammography screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mammography screening only (No Intervention): This group will receive their standard of care mammogram only. Participants in this arm will not receive the FAST MRI.
  Participants will complete 4 questionnaires at 3 time points: enrollment; 2 weeks after they receive their mammogram; 6 months after their mammogram.
- FAST MRI and mammogram screening (Experimental): Patients in this group will receive Breast MRI and annual mammography. Participants will complete 4 questionnaires at 3 time points: enrollment; 2 weeks after they receive their mammogram; 6 months after their mammogram. The intervention is the addition of the FAST Breast MRI.
  Interventions: Other: FAST MRI and mammography screening

INTERVENTIONS:
Other: FAST MRI and mammography screening — Patients in this group will receive Breast MRI and annual mammography. Participants will complete 4 questionnaires at 3 time points: enrollment; 2 weeks after they receive their mammogram; 6 months after their mammogram.
  Other Names: FAST MRI
  Arms: FAST MRI and mammogram screening

SUMMARY:
Breast Magnetic Resonance Imaging (MRI) has been shown to be the most accurate test for detecting breast cancer however, MRI is not always reliable because it can indicate the presence of cancer when in reality, there is none; this is called a 'false positive' result. A history of breast carcinoma alone does not qualify a patient for ongoing monitoring with breast MRI. This study is being done to assess a new technique called FAST breast MRI. A FAST breast MRI is different than a traditional breast MRI because it has much fewer sequences and takes approximately 3 minutes for the scan. MRI sequences are combinations of magnetic pulses that collect information about the tissues. There is no radiation associated with an MRI.

The purpose of this study is to determine the impact on patient health when a FAST breast MRI is used as a screening technique in women with a personal history of cancer. It has been shown that FAST breast MRI is similar to routine breast MRI in the detection of breast cancer, but it has not been proven that FAST breast MRI will help women who have a personal history for breast cancer. Currently, routine breast MRI is not part of the standard of care in screening for breast cancer in women who have a prior personal history of breast cancer. By evaluating FAST MRI the investigators are able to study the effects of this short MRI on cancer detection in women with a personal history of breast cancer, and on the impact on overall health. The investigators estimate that 300 participants will be enrolled in the study from The Ottawa Hospital Cancer Centre at The Ottawa Hospital, General Campus and the Women's Breast Health Centre at The Ottawa Hospital, Civic Campus. All of the participants have had a history of breast carcinoma.

DETAILED DESCRIPTION:
Given the demand for breast MRI screening by breast cancer survivors and oncologists, we plan to perform a randomized controlled trial in a select patient population of breast cancer survivors who would not normally be eligible for breast MRI screening. This study will determine whether using FAST MRI in addition to mammography will reduce anxiety in patients compared to the current standard of care: mammography alone. If it turns out to reduce anxiety, the next step would be to conduct a large-scale multi-centre randomized control trial (RCT) to evaluate whether FAST MRI is more sensitive and whether the increased sensitivity leads to improved clinical outcomes.

The purpose of our study is to determine the impact on patient anxiety of FAST Breast MRI as a surveillance technique in women with a personal history of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* English or French speaking female patients over the age of 18 years, with a personal history of a diagnosis of breast carcinoma (including ductal carcinoma in situ (DCIS) and invasive ductal or lobular carcinoma) within the past 10 years.
* Patients must have completed treatment for their breast cancer.
* Moderate risk for recurrence of breast cancer, defined as lifetime risk of breast cancer greater than 12% (average risk) and less than 25% (high risk) as defined using the Breast and Ovarian Analysis of Disease Incidence and Carrier Estimation Algorithm (BOADICEA) model (see Appendix A)
* Patients who have undergone unilateral mastectomy or breast conservation surgery.
* Normal renal function: estimated glomerular filtration rate (eGFR) > 30 ml/min/m2

Exclusion Criteria:

* Patients unable to undergo an MRI, due to either physical or mental issues (i.e.: anxiety or severe claustrophobia). Also, patient with a known allergy to gadolinium, or severe renal failure will be excluded.
* Pregnant or breastfeeding patients.
* Patients who have had a breast MRI within the last 6 months.
* Patients already receiving high-risk breast MRI screening, such as the Ontario Breast Screening Program (OBSP) high-risk program and the Women's Breast Health Center (WBHC) high-risk program.
* Patients who have undergone bilateral mastectomies.
* Poor renal function: estimated glomerular filtration rate (eGFR) < 30 ml/min/m2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-10; Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with reduced anxiety as a result of having a FAST MRI | up to 12 months

SECONDARY OUTCOMES:
Numbers of recurrent tumors in each arm | 12 months

OTHER OUTCOMES:
Number of tumors missed by mammography | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Seely, MD FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Planning on submitting preliminary results to RSNA 2017 and full publication by Oct 2018.

REFERENCES:
- [Derived] Fonseca MM, Alhassan T, Nisha Y, Koszycki D, Schwarz BA, Segal R, Arnaout A, Ramsay T, Lau J, Seely JM. Randomized trial of surveillance with abbreviated MRI in women with a personal history of breast cancer- impact on patient anxiety and cancer detection. BMC Cancer. 2022 Jul 15;22(1):774. doi: 10.1186/s12885-022-09792-x. PMID 35840916